CLINICAL TRIAL: NCT03785353
Title: The Effects of Pain Neuroscience Education in a Spanish-Speaking Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenandoah University (Other)
Responsible Party: Principal Investigator, Aaron Hartstein, Assistant Professor of Physical Therapy, Shenandoah University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ShenandoahU(2018-2019)
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Pain; Educational Problems
Keywords: Pain Neuroscience Education; Spanish-speaking
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Participants will arrive at a location TBD on the day of data collection. Consent forms will be dispersed to participants, who will be able to ask any questions they may have before signing. A Spanish-speaking researcher will be available to answer those questions. After consent is received, each participant will draw a random number that will be used to link their responses to pre- and post-lecture surveys. After consent is received, a pre-test on pain knowledge and beliefs will be administered. A 30-minute Pain Neuroscience Education (PNE) lecture will be given to participants in Spanish. A post-test on pain knowledge and beliefs will be administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PNE Group (Experimental): A group of Spanish-speaking individuals will listen to a translated lecture related to PNE (PNE lecture). They will fill out the R-NPQ pre and post the lecture.
  Interventions: Behavioral: PNE lecture

INTERVENTIONS:
Behavioral: PNE lecture — A translated (from English to Spanish) lecture on Pain Neuroscience Education

SUMMARY:
Pain Neuroscience Education (PNE) has been shown to be effective to alter beliefs and decrease pain among individuals with musculoskeletal pain. Additionally, PNE has been shown to alter beliefs among middle school children. This study plans to assess the effects of PNE within a group of Spanish-speaking individuals.

DETAILED DESCRIPTION:
Chronic pain is a topic of discussion that is becoming increasingly prevalent among healthcare professionals. With the ever-growing opioid epidemic, there are a variety of discussions on different modes of treatment other than opioid prescription. Pain neuroscience education, or PNE, is one of these alternative treatment options. PNE focuses on a patient's understanding of pain itself and relates this to the current pain they are experiencing. PNE is often a discussion between provider and patient that utilizes a series of stories, metaphors, and examples where pain is described from a point of view that is not strictly medical. Recent literature suggests there is a lack of knowledge regarding pain in the United States, particularly in the Spanish-speaking population. This population is also less likely to seek a physician's advice for pain management. For these reasons, this study will focus on the Spanish-speaking population within the Winchester community. Due to success within prior PNE studies, this study will be conducted through a classroom lecture. The overarching purpose of this study is to examine the change in knowledge of pain in the Spanish-speaking population immediately following a PNE lecture composed of stories, metaphors, and examples about pain. Because Spanish-speaking individuals are less likely to seek out a medical provider, the study may support an additional treatment option for managing chronic pain. Not only will this provide further research to support the benefits of PNE, but there is the potential to modify a participant's perception of their own pain through this educational lecture.

ELIGIBILITY:
Inclusion Criteria:

* Participants must speak Spanish at least 50% of the time at home OR Spanish must be the first language learned. Participants must also be willing to sit and listen to lecture and fill out quiz before and after.

Exclusion Criteria:

* Any individual under the age of 18 will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
R-NPQ | Immediately post-lecture
  Revised Neuroscience of Pain Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sheri A Hale, PT, PhD, ATC, Study Director — Shenandoah University
Locations (1):
- Shenandoah University, Winchester, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Louw A, Podalak J, Zimney K, Schmidt S, Puentedura EJ. Can pain beliefs change in middle school students? A study of the effectiveness of pain neuroscience education. Physiother Theory Pract. 2018 Jul;34(7):542-550. doi: 10.1080/09593985.2017.1423142. Epub 2018 Jan 8. PMID 29308954
- [Result] Louw A, Zimney K, Puentedura EJ, Diener I. The efficacy of pain neuroscience education on musculoskeletal pain: A systematic review of the literature. Physiother Theory Pract. 2016 Jul;32(5):332-55. doi: 10.1080/09593985.2016.1194646. Epub 2016 Jun 28. PMID 27351541
- [Result] Louw A, Zimney K, O'Hotto C, Hilton S. The clinical application of teaching people about pain. Physiother Theory Pract. 2016 Jul;32(5):385-95. doi: 10.1080/09593985.2016.1194652. Epub 2016 Jun 28. PMID 27351903